CLINICAL TRIAL: NCT00062855
Title: Phase I Study of Chemokine and Cytokine Gene Modified Autologous Neuroblastoma Cells for Treatment of Relapsed/Refractory Neuroblastoma Using an Adenoviral Vector (CYCHE)
Brief Title: Using Gene Modified Neuroblastoma Cells for the Treatment of Relapsed/Refractory Neuroblastoma
Acronym: CYCHE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Malcolm Brenner, Professor, Director Center for Cell and Gene Therapy, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H6442; Cyche; NCT00002713 (obsolete NCT alias)
Record Dates: First submitted 2003-06-17; First posted 2003-06-18 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Neuroblastoma
Keywords: GENE MODIFIED AUTOLOGOUS NEUROBLASTOMA CELLS; Gene Therapy
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gene Modified Neuroblastoma Cells (Experimental): Gene modified neuroblastoma cells given as 4 subcutaneous injections over 5 weeks
  Interventions: Procedure: Skin Biopsy; Genetic: Gene Modified Neuroblastoma Cells

INTERVENTIONS:
Procedure: Skin Biopsy
Genetic: Gene Modified Neuroblastoma Cells — The first two injections will be given at week 1 and week 2 (i.e., separated by one week). Patients will then have a two-week rest and the remaining two injections will be given (again separated by one week) at week 4 and week 5.
  A complete evaluation for evidence of toxicity and response will be performed at week 8 (after a 3 week rest).
  At the 8 week (month 2) evaluation, in the absence of progressive disease requiring therapy without excessive toxicity and if more transduced cells are available, the patient will have the option to receive four additional SC injections each separated by 1 month at the higher of the two dosage levels they originally received.

SUMMARY:
This research study is designed to determine the safety and dosage of special cells that may make a patients own immune system fight the cancer. To do this we will put two special genes into cancer cells taken from the patients body. The genes we put in make the cancer cells produce lymphotactin, a natural substance that attracts immune system cells to the cancer, and IL-2 a natural substance that may help the immune system kill cancer cells. Some of these cells will then be put back in the patient's body. Studies of cancers in animals and in cancer cells that are grown in laboratories suggest that substances like lymphotactin and IL-2 help the body kill cancer cells. A treatment similar to this has been used in ten children previously and similar treatments are being used in adults with other cancers.

The purpose of this study is to learn the side effects and safe 'dosage' of these special cells.

DETAILED DESCRIPTION:
Neuroblastoma cells taken from the patient will be separated in the laboratory and two specially produced human viruses (adenovirus) that carry the lymphotactin and the IL-2 gene were put into the cells. These lymphotactin and IL-2 genes are meant to help the immune system fight the cancer.

The modified cancer cells will be injected under the patient's skin. There will be four shots. The second and subsequent shots will have ten times as many cells producing lymphotactin as the first. We do not know the best amount of special cells to use, so different patients will get different numbers of cells.

Before the second shot, and then again about 2 weeks later, we will remove some of the modified cells from the patient's body and study them. We will do this by removing a section of skin (referred to as a skin biopsy) at the place where the cells were injected. This test will help us to see whether or not the modified cells are killing cancer cells.

To study how the immunity is working in the patient's system, we will take blood samples prior to each injection, two to four days after each injection, and may repeat this 5-7 days after each injection if your doctor thinks that is necessary.

After patients have received the first set of 4 injections a complete evaluation is performed to see how this research treatment is working. If these evaluations look okay and if more injections are available, patients will have the option to receive a second set of 4 injections. If patients receive the second set of 4 injections, they will again have blood samples taken after each injection.

After injections stop, all patients will have blood samples collected once a month for a year, and then once a year for fifteen years.

To see if this research treatment is working, we will do CAT scans, MRIs, or bone scans (these are different types of x-rays). We will also take a bone marrow biopsy (bone marrow will be removed by use of a needle so that it can be looked at under the microscope). These tests will be done prior to treatment and again eight weeks later. In addition, if patients receive the second set of four injections, these tests will be repeated at six months.

ELIGIBILITY:
* All patients under 21 years of age at diagnosis with recurrent, advanced stage neuroblastoma.
* Patients must have a life expectancy of at least 8 weeks.
* Patients must have recovered from the toxic effects of all prior chemotherapy before entering this study, and have an absolute lymphocyte and neutrophil count of >500/mm3 each.
* Patients must not be currently receiving any investigational agents or have not received any tumor vaccines within the previous six weeks.
* Patients must not be HIV-positive.
* Patients must have bilirubin <1.5 mg%.
* Patients must have creatinine <1.5 mg/dl.
* Patients must have ECOG performance status of 0-2.
* Patients must have autologous transduced neuroblastoma cells available that are demonstrably producing >150 pg IL-2/106 cells/24 hr and are secreting Lptn.
* Patients or legal guardians must sign an informed consent indicating that they are aware this is a research study and have been told of its possible benefits and toxic side effects. Patients or their guardians will be given a copy of the consent form.
* Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 3 months after the study is concluded. The male partner should use a condom.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 1997-11; Primary Completion 2001-08 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
To determine the safety of up to four subcutaneous (SC) injections of autologous neuroblastoma cells which have been genetically modified by adenoviral vectors to secrete lymphotactin (Lptn) and Interleukin-2 (IL-2). | 2 months
To determine the safety of up to eight (total) of these injections in patients who have received the first four injections without unacceptable toxicity and have evidence of stable disease or better after receiving these injections. | 6 months

SECONDARY OUTCOMES:
To determine whether MHC restricted or unrestricted antitumor immune responses are induced by SC injection of modified autologous neuroblasts and the cell doses required to produce these effects. | 3 weeks
To obtain preliminary data on the antitumor effects of this treatment regimen | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Brenner, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States